CLINICAL TRIAL: NCT01904812
Title: Longitudinal Study of Quality of Life and Activity in Systemic Lupus Erythematosus
Acronym: EQUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Besancenot PHRC N 2010
Record Dates: First submitted 2013-07-12; First posted 2013-07-22 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2013-07

CONDITIONS: Lupus Erythematosus

ARMS (1):
- Lupus erythematosus (Other)
  Interventions: Other: Questionnaire about quality of life and satisfaction

INTERVENTIONS:
Other: Questionnaire about quality of life and satisfaction

SUMMARY:
Systemic lupus erythematosus is a complex disease whose evaluation in everyday practice and in clinical research requires several aspects to be taken into account, in particular the impact of disease activity on quality of life. To date, the effect of systemic lupus on quality of life has only been described using generic questionnaires. Among the specific questionnaires for systemic lupus, the LupusQol, which has been validated in French, shows interesting psychometric properties. The determinants of quality of life specifically related to the disease are still unknown and could be studied using a longitudinal cohort thanks to the French version of the LupusQol.

ELIGIBILITY:
Inclusion Criteria:

* - Patients meeting ACR 1997 classification criteria for systemic lupus erythematosus.
* Patients able to understand written and spoken French.
* Patients aged from 18 to 75 years
* Patients who have received written and oral information about the research.

Exclusion Criteria:

* - Patients aged less than 18 years
* Patients aged more than 75 years
* Severe mental retardation Any impairment of abilities to understand that make self-evaluation impossible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
data for quality of life and satisfaction | participants will be followed for the duration of hospital stay, an expected average of 3 months
  Quality of life and satisfaction will be evaluate by questionnaire as Questionnaire SLEQOL, QUESTIONNAIRE LUPUSQOL, QUESTIONNAIRE MFI-20

SECONDARY OUTCOMES:
Clinical data | participants will be followed for the duration of hospital stay, an expected average of 3 months
  Question about any recent hospitalization pregnancy contraception Compliance score of Girerd Fatigue score MFI-20 tobacco consumption Score of CES-D depression Score stress response WCC

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François BESANCENOT, Principal Investigator — CHU Dijon - Department of Internal Medicine and Systemic Diseases
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Derived] Thibault T, Bourredjem A, Maurier F, Wahl D, Muller G, Aumaitre O, Seve P, Blaison G, Pennaforte JL, Martin T, Magy-Bertrand N, Audia S, Arnaud L, Amoura Z, Devilliers H; EQUAL Study Group. The mediating effect of fatigue in impaired quality of life in systemic lupus erythematosus: mediation analysis of the French EQUAL cohort. Rheumatology (Oxford). 2023 Sep 1;62(9):3051-3058. doi: 10.1093/rheumatology/kead020. PMID 36655762
- [Derived] Corneloup M, Maurier F, Wahl D, Muller G, Aumaitre O, Seve P, Blaison G, Pennaforte JL, Martin T, Magy-Bertrand N, Berthier S, Arnaud L, Bourredjem A, Amoura Z, Devilliers H; EQUAL Study Group. Disease-specific quality of life following a flare in systemic lupus erythematosus: an item response theory analysis of the French EQUAL cohort. Rheumatology (Oxford). 2020 Jun 1;59(6):1398-1406. doi: 10.1093/rheumatology/kez451. PMID 31620787